CLINICAL TRIAL: NCT00862082
Title: A Randomized Phase I/II, Multi-Center, Open-Label Trial of PR104 and Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Randomized Phase 1/2 Open-Label Trial of PR104 and Sorafenib in Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PR104 plus sorafenib was poorly tolerated in patients with advanced HCC
Sponsor: Proacta, Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR104-2002; NCT00838604 (obsolete NCT alias)
Record Dates: First submitted 2009-03-12; First posted 2009-03-16 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — PR-104; Sorafenib

ARMS (1):
- PR104 + Sorafenib (Experimental): PR104 will be administered IV once every four weeks, in addition to 400mg sorafenib PO twice daily
  Interventions: Drug: PR104 550 mg/m^2 + sorafenib; Drug: PR104 770 mg/m^2 + sorafenib

INTERVENTIONS:
Drug: PR104 550 mg/m^2 + sorafenib — 550 mg/m^2 PR104 IV on day 1 of each 28 day cycle + 400 mg sorafenib PO twice daily. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: PR-104; Nexavar
Drug: PR104 770 mg/m^2 + sorafenib — 770 mg/m^2 PR104 IV on day 1 of each 28 day cycle + 400 mg sorafenib PO twice daily. Number of Cycles: until progression or unacceptable toxicity develops.
  Other Names: PR-104; Nexavar

SUMMARY:
The current understanding of PR104 justifies the evaluation of PR104 with sorafenib in patients with hepatocellular carcinoma. These include:

* Hypoxia. Hepatocellular Carcinoma (HCC) is likely to demonstrate a level of hypoxia sufficient to activate PR104 to its active metabolites PR104H and PR104M. In addition, in preclinical models, sorafenib has been demonstrated to increase the degree of hypoxia in tumors following treatment.
* Non-overlapping toxicity. PR104 and sorafenib do not share major toxicities. It is anticipated that both drugs can be administered at their full single agent dose when used in combination.
* Aldo-keto reductase 1C3 (AKR1C3). HCC has been shown to express high levels of AKR1C3 which should lead to selective activation of PR104 within both hypoxic and oxic HCC cells.
* Preclinical data. The use of sorafenib and PR104 alone and in combination in a hepatocellular carcinoma model demonstrates activity of PR104 as a single agent and increased activity when PR104 and sorafenib are used in combination.

The current study will provide an estimate of the activity of PR104 in subjects with HCC. This information will prove valuable in defining the future clinical development of PR104, and in determining if PR104 has sufficient activity in HCC to warrant a larger phase III registration study in this indication.

Primary objectives

* Phase I: Determine the maximum tolerated dose (MTD) of PR104 when used in combination with standard dose sorafenib
* Phase II: Estimate the response rate (RR) of PR104/sorafenib [Note: Phase II was never initiated]

Secondary objectives

* Evaluate survival
* Evaluate Progression Free Survival (PFS)
* Evaluate time to progression (TTP)
* Evaluate safety
* Evaluate the pharmacokinetics (PK) of sorafenib, PR104 and PR104 metabolites
* Collect diagnostic biopsy samples for the determination of aldo-keto reductase 1C3
* Collect plasma samples for assessment of potential biomarkers of tumor hypoxia

DETAILED DESCRIPTION:
A randomized phase I/II, multi-center, open-label, study with a single arm phase I portion to determine the appropriate dose of PR104 combined with sorafenib, followed by a phase II portion with randomization between sorafenib and sorafenib/PR104.

Following informed consent, subjects will undergo baseline evaluation with history, physical exams, blood work and disease assessment. Selected subjects will undergo PK assessment of sorafenib, PR104 and PR104 metabolites.

In the phase I portion of the study, the starting dose of PR104 will be 770 mg/mg2 in combination with standard dose sorafenib. PR104 will be administered on an every 4 week schedule with the dose of PR104 escalated in a standard phase I fashion (3 subjects per cohort, dose escalation between cohorts) in order to determine the MTD of PR104. Cohorts may be expanded up to 12 subjects to better define toxicity at a particular dose level. Following determination of the MTD of PR104, new subjects will be entered into the phase II portion of the study. [Note: the Phase II portion was never initiated]

In the phase II portion of the study, subjects will be randomized between sorafenib, 400 mg, by mouth (PO), twice a day (the approved dose and schedule) versus sorafenib with PR104 at the dose determined in the phase I portion of the study. PR104 will be administered every 4 weeks (one cycle). Subjects will be evaluated each week during cycle 1 and every two weeks thereafter. A disease assessment will be performed after every two cycles. Subjects with progression will be removed from study. Subjects with a response or stable disease may continue on study if this is considered beneficial by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Advanced-stage hepatocellular carcinoma considered non-operable that is suitable for treatment with sorafenib. Subjects who have demonstrated progression following initial surgical or locoregional therapy are eligible
* Confirmed hepatocellular carcinoma by pathological analysis (tissue aspirate or biopsy)
* No previous systemic therapy for hepatocellular carcinoma
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Child-Pugh liver function class A
* Life expectancy of 12 weeks or more
* Adequate hematologic function [Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L; platelet count ≥100×10^9 per liter; hemoglobin ≥8.5 g per deciliter maintained in the absence of red blood cell transfusions; and prothrombin time international normalized ratio ≤1.7; or prothrombin time ≤2 seconds above control]
* Adequate hepatic function (albumin ≥2.8 g per deciliter; total bilirubin ≤2 mg per deciliter [51.3 μmol per liter]; and alanine aminotransferase and aspartate aminotransferase ≤5 times the upper limit of the normal range)
* Adequate renal function (serum creatinine ≤1.5 times the upper limit of the normal range or creatinine clearance ≥60 mL/min).
* At least one untreated target lesion that could be measured in one dimension, according to the Response Evaluation Criteria in Solid Tumors (RECIST)
* Concomitant systemic antiviral therapy allowed

Exclusion Criteria:

* Previous molecularly targeted therapies or any other systemic treatment for hepatocellular carcinoma
* Active concomitant malignancy likely to effect any of the primary or secondary outcome measures in the current study
* Women who are pregnant, breast-feeding or planning to become pregnant during the study
* Men or women of reproductive-potential who are unwilling to use an effective method of contraception during the study and for 30 days following the last dose of study medication
* Evidence of a significant medical disorder or laboratory finding that, in the opinion of the Investigator, compromises the subject's safety during study participation such as: uncontrolled infection or infection requiring a concomitant parenteral antibiotic; uncontrolled diabetes; congestive heart failure; myocardial infarction within 6 months of study; chronic renal disease; or coagulopathy (excluding prophylactic anticoagulation)
* Active central nervous system metastatic disease requiring intervention
* Less than four weeks since major surgery
* Known Human Immunodeficiency Virus (HIV) positivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2010-01 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - University of Arizona, Tucson, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - University of California, Irvine, Orange, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Pacific Oncology/Hematology, San Francisco, California
  - Northwestern University, Chicago, Illinois
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Columbia University Medical Center, New York, New York
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong
- Singapore General Hospital, Singapore, Singapore
- Taiwan (6):
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center, Liouying, Tainan
  - Cathay General Hospital, Taipei
  - National Taiwan University Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Groups:
- PR104 550 mg/m^2 + Sorafenib: 550 mg/m^2 PR104 administered IV every 4 weeks + Standard dose sorafenib (400 mg PO twice daily)
- PR104 770 mg/m^2 + Sorafenib: 770 mg/m^2 PR104 administered IV every 4 weeks + Standard dose sorafenib (400 mg PO twice daily)
Period: Overall Study
Arm/Group | PR104 550 mg/m^2 + Sorafenib | PR104 770 mg/m^2 + Sorafenib
Started | 8 | 6
Completed | 3 | 5
Not Completed | 5 | 1
Not completed — Sponsor decision to terminate the study | 5 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PR104 550 mg/m^2 + Sorafenib | PR104 770 mg/m^2 + Sorafenib | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (13) | 59 (13) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
  Taiwan | 5 | 2 | 7
  Hong Kong | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of PR104 When Used in Combination With Standard Dose Sorafenib in the Phase I Population
Time Frame: 4 weeks (1 cycle)
Measure: Number; unit: mg/m2
Groups:
- Cohorts 1 and 2: 770 and 550 mg/m^2 PR104 administered IV every 4 weeks + Standard dose sorafenib (400 mg PO twice daily)
Arm/Group | Cohorts 1 and 2
Number analyzed (Participants) | 14
mg/m2 | NA — There were no DLTs, however myelosuppression in several patients led to the decision to discontinue the study; therefore, a MTD was not determined.

2. Secondary Outcome: Safety and Tolerability: Serious Adverse Events
Description: The number of participants with at least one Serious Adverse Event was measured.
Time Frame: 30 days following the last administration of study treatment
Measure: Number; unit: participants
Groups:
- Cohort 1: 770 mg/m^2 PR104 administered IV every 4 weeks + Standard dose sorafenib (400 mg PO twice daily)
- Cohort 2: 550 mg/m^2 PR104 administered IV every 4 weeks + Standard dose sorafenib (400 mg PO twice daily)
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 6 | 8
participants | 2 | 5

3. Secondary Outcome: Pharmacokinetics [Maximum Plasma Concentration (Cmax)] of PR104 and PR104 Metabolites in Cohort 1 (770 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in pharmacokinetic (PK) sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- PR104A; PR104G: major plasma metabolite
- PR104S1: semi-mustard metabolite
- PR104H; PR104M: activated reduced metabolites
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
ng/ml
  Cmax Cycle 1 | 7.1 (3.2) | 7.6 (1.9) | 9.6 (2.3) | 0.17 (0.15) | 0.21 (0.11) | 0.04 (0.02)
  Cmax Cycle 2 | 6.0 (3.3) | 7.6 (1.0) | 10.4 (2.2) | 0.18 (0.07) | 0.20 (0.05) | 0.04 (0.02)

4. Secondary Outcome: Pharmacokinetics [Half Life (T1/2)] of PR104 and PR104 Metabolites in Cohort 1 (770 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in PK sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
hr
  T1/2 Cycle 1 | 0.15 (0.10) | 0.75 (0.35) | 0.62 (0.08) | 0.87 (0.11) | 1.37 (0.18) | 3.57 (0.82)
  T1/2 Cycle 2 | 0.17 (0.11) | 0.85 (0.20) | 0.67 (0.17) | 0.79 (0.14) | 1.05 (0.35) | 02.93 (2.48)

5. Secondary Outcome: Pharmacokinetics [Area Under the Curve(AUC)] of PR104 and PR104 Metabolites in Cohort 1 (770 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in PK sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2
ng.h/ml
  AUC Cycle 1 | 5.1 (3.2) | 11.0 (4.4) | 12.3 (1.3) | 0.26 (0.23) | 0.47 (0.27) | 0.22 (0.09)
  AUC Cycle 2 | 4.3 (2.9) | 10.6 (0.1) | 15.8 (2.9) | 0.28 (0.10) | 0.42 (0.04) | 0.19 (0.17)

6. Secondary Outcome: Pharmacokinetics (Cmax) of PR104 and PR104 Metabolites in Cohort 2 (550 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in PK sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 5 | 5 | 1 | 5 | 5 | 5
ng/ml
  Cmax Cycle 1 | 3.2 (1.1) | 15.8 (8.9) | 4.9 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle | 0.21 (0.18) | 0.72 (0.80) | 0.12 (0.12)
  Cmax Cycle 2 | 4.3 (0.7) | 14.6 (10.4) | 5.8 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle. | 0.17 (0.17) | 0.69 (0.78) | 0.16 (0.13)

7. Secondary Outcome: Pharmacokinetics (T1/2) of PR104 and PR104 Metabolites in Cohort 2 (550 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in PK sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 5 | 5 | 1 | 5 | 5 | 5
hr
  T1/2 Cycle 1 | 0.10 (0.01) | 0.68 (0.04) | 0.53 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle. | 0.69 (0.20) | 0.84 (0.34) | 1.02 (0.42)
  T1/2 Cycle 2 | 0.09 (0.01) | 0.79 (0.23) | 0.50 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle. | 0.90 (0.44) | 0.91 (0.25) | 0.99 (0.52)

8. Secondary Outcome: Pharmacokinetics (AUC) of PR104 and PR104 Metabolites in Cohort 2 (550 mg/m^2 Dose Group)
Time Frame: Day 1 of Cycles 1 and 2
Population: Participation in PK sampling was optional to subjects, therefore not all subjects in the study were analyzed.
Measure: Mean (Standard Deviation); unit: ng.h/ml
Arm/Group | PR104 | PR104A | PR104G | PR104S1 | PR104H | PR104M
Number analyzed (Participants) | 5 | 5 | 1 | 5 | 5 | 5
ng.h/ml
  AUC Cycle 1 | 2.4 (0.8) | 19.7 (9.7) | 6.4 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle. | 0.30 (0.23) | 0.81 (0.71) | 0.18 (0.13)
  AUC Cycle 2 | 3.3 (0.6) | 22.7 (18.2) | 7.6 (NA) — Not determined for PR-104G due to the availability of only one subject's dataset from each cycle. | 0.31 (0.21) | 1.07 (1.02) | 0.25 (0.18)

ADVERSE EVENTS:
Arm/Group | PR104 550 mg/m^2 + Sorafenib | PR104 770 mg/m^2 + Sorafenib
Serious Adverse Events (participants affected / at risk) | 5/8 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PR104 550 mg/m^2 + Sorafenib (N=8) | PR104 770 mg/m^2 + Sorafenib (N=6)
Abdominal Pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Decrease in general condition (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Fever in absence of neutropenia (General disorders) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PR104 550 mg/m^2 + Sorafenib (N=8) | PR104 770 mg/m^2 + Sorafenib (N=6)
Leukopenia (Blood and lymphatic system disorders) | 7 | 4
Anemia (Blood and lymphatic system disorders) | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 6 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 5
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1
Fatigue (General disorders) | 3 | 3
Induration (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 3
Alanine aminotransferase increased (Investigations) | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 3 | 1
International normalised ratio increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Diarrhea (Gastrointestinal disorders) | 3 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 2
Leukocytoclastic vasulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 3 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Phase II part of study never initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Single site data may be published/presented prior to the publication of multi-center data from overall study if agreed to by the sponsor in writing, or 12 months have elapsed following termination or completion of the study, whichever comes first.